CLINICAL TRIAL: NCT02265042
Title: Effect of Electrostimulation on Denervated Muscles in Individuals With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Principal Investigator, Bersch-Porada Ines, PhD in Medical Sciences, Swiss Paraplegic Research, Nottwil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-13
Record Dates: First submitted 2014-10-07; First posted 2014-10-15 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- electrical stimulation (Experimental): electrical Stimulation using the Stimulette device
  Interventions: Device: Stimulette

INTERVENTIONS:
Device: Stimulette — electrical stimulation device by Dr. Schuhfried Medizintechnik GmbH, Vienna, Austria

SUMMARY:
The aim of the study is to investigate whether there is an effect of electrical stimulation on the denervated gluteus muscle (buttocks) in individuals with chronic spinal cord injury. The expected outcome is an increase in muscle volume and a better pressure distribution during sitting. The stimulation of the gluteus muscle is performed daily for 35 minutes over a period of six months. The muscle volume and the pressure distribution are measured before stimulation, three months after having started stimulation and after six months.

ELIGIBILITY:
Inclusion Criteria:

* chronic spinal cord injury (min. 2 years after injury)
* lesion height from T10-L5
* ASIA (American Spinal Cord Injury Association) Impairment Scale A

Exclusion Criteria:

* acute pressure sore in stimulated area (M. gluteus)
* arteriosclerosis
* skin irritation or infection in stimulated area (M. gluteus)
* < 3 months after plastic surgery in stimulated area (M. gluteus)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
change in muscle volume | day 0 to 3 months
  determination of muscle volume using magnetic resonance images

SECONDARY OUTCOMES:
change in muscle volume | 3 months to 6 months
  determination of muscle volume using magnetic resonance images
change in sitting pressure | day 0 to 3 months
  pressure mapping system
change in sitting pressure | 3 months to 6 months
  pressure mapping system
change in quality of life | day 0 to 3months
  questionnaire
change in quality of life | 3 months to 6 months
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland